CLINICAL TRIAL: NCT02032940
Title: Non-Enhanced Magnetic Resonance Angiography With the t-SLIP Technique
Acronym: MRAtSLIP
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Miami Cardiac and Vascular Institute (Other)
Responsible Party: Principal Investigator, Constantino Pena, MD, Constantino Pena, MD. Medical Director of Vascular Imaging, Miami Cardiac and Vascular Institute
Other Study IDs: 2013-020
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Focus of Study is MRI
Keywords: MRI, Angiography, Pulse Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard Sequence Imaging MRI: Patients requiring MRI. All Comers accepting study participation.
- Additional Pulse Sequence Increased: Patients requiring MRI. All comers accepting study participation and the run of additional pulse sequences during MRI procedure.

SUMMARY:
The purpose of the study is to create MR images using an investigative technique called pulse sequences with new computer software programs. The sequence will allow us to image vessels without injecting contrast agents.

DETAILED DESCRIPTION:
The t-SLIP Investigational Study Sequences are designed to compare t-SLIP to standard MR contrast enhanced imaging techniques to establish the diagnosic benefits of t-SLIP compared to contrast enhanced MR techniques. The t-SLIP Investigational Study Sequences will be used for vascular MRI Imaging including, but no limited to, MRA of the renal, mesenteric, abdominal aortic, iliac and femoral arteries. We will be targeting all adult patients undergoing standard body MRA examinations without anesthesia.

The time spatial labeling inversion pulse (t-SLIP) technique is used for non contrast enhanced MR angiography imaging. It produces bright blood spin labeling images by using a single acquisition with a combination of a spatially nonselective inversion pulse and a spatially selective inversion pulse. The nonselective pulse inverts the magnetization of the entire imaging area. The spatially selective pulse, applied upstream of the arteries of interest, reverts those protons to full magnetization. A pre defined time delay between tagging and imaging allows the tagged spins to reach the imaging region and suppresses background tissue within the imaging region to some extent.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are considered candidates and scheduled for standard contrast enhanced MRA can be included in the study.

Exclusion Criteria:

* Patients that can not undergo standard MRA

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Patients Needing Thoracic, Aortic, Renal, Iliac and/or Femoral Vasculature MRIs
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Degree of enhancement by evaluation of the Thoracic, Aortic, Renal, Iliac and Femoral Vasculature Images | 2 Years
  The project proposal is to acquire the additional sequence as part of the standard examination and then to compare the sequence to the standard MR contrast enhanced imaging techniques in order to establish the diagnostic benefits of this sequence compared to contrast enhanced MR techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Constantino Pena, MD, Principal Investigator — Baptist Cardiac and Vascular Institute
Locations (2):
- United States (2):
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Miami Cardiac and Vascular Institute, Miami, Florida

IPD SHARING:
Plan to Share IPD: No